CLINICAL TRIAL: NCT04117204
Title: Identifying a Cardiorenal Protective Diet in a Lower-income African American Population With Chronic Kidney Disease at Risk for Cardiovascular Disease.
Brief Title: Cardiorenal Protective Diet
Acronym: CPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 018-095
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Hypertension
Keywords: CVD; Dietary Intervention
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hypertension | interventions — Fruit; Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruits and Vegetables (Experimental): This group will receive a prescribed amount of free fruits and vegetables (F&V) for 6 weeks of pick-up at a farm stand or direct delivery. After 6 weekly pick-up/deliveries, participants will be provided vouchers and reminders to obtain F&V at farm stands for an additional 6 weeks with minimal contact.
  Interventions: Other: Fruits and Vegetables
- Wait List Control (No Intervention): This group will not receive a prescribed amount of free fruits and vegetables (F&V) for 12 weeks. They will serve as the control group. After 12 weeks of control and data comparisons, they will be given 12 weeks of vouchers with minimal contact.

INTERVENTIONS:
Other: Fruits and Vegetables — Fruits and Vegetable delivery, once a week for 12 weeks.
  Arms: Fruits and Vegetables

SUMMARY:
This study will evaluate providing fruits and vegetables in a sustainable community care clinic setting, in addition to routine medical care, to individuals with CKD (Stage 2-4) on CKD and CVD risk, or cardio-renal risk factors. Further, metabolomics profiling will be used to study how change in the diet affects disease risk. Data from this study will be published in peer-reviewed journals, presented at national conferences, and will serve as pilot data to guide and strengthen applications for NIH funding.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in a 3-month F&V study.
* Positive urine dipstick (Proteinuria and/or Albumin-to-Creatinine Ratio >=10).
* African-American (self-declared) race
* A current diagnosis of hypertension or a current blood pressure reading consistent with hypertension (SBP >= 140 and/or DBP >=90).
* Access to the internet via personal computer or mobile device.
* Ability to read and write in English.

Exclusion Criteria:

* Negative urine dipstick.
* Currently receiving dialysis or needing dialysis (Stage 5 Kidney Disease)
* Have received or need a kidney transplant.
* Pregnant or planning to become pregnant in the next 6 months.
* Baseline urine potassium > 60mEq/g creatinine
* Negative diagnosis of hypertension or blood pressure reading (SBP <140 or DBP <90).
* Nephrotic proteinuria demonstrated on urine ACR measurement.
* Lacking access to the internet via personal computer or mobile device.
* Unable to read or write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in fruit and vegetable intake at 6 weeks and 3 months. | Baseline; 6 weeks and 3 months
  Track changes in fruit and vegetable intake via ASA24 dietary recall food diary.
Changes from baseline in systolic and diastolic blood pressure at 6 weeks and 3 months. | Baseline; 6 weeks and 3 months
  Measure changes in systolic/diastolic blood pressure (mmHg) to assess cardiovascular disease (CVD) risk.
Change from baseline of urine albumin-to-creatinine ration (ACR) at 6 weeks and 3 months. | Baseline; 6 weeks and 3 months
  Measure of renal damage.

SECONDARY OUTCOMES:
Metabolomics will be used to profile how changes in diet effects disease risk. | Baseline and 6 Weeks
  Urine and plasma specimens will be collected for metabolomic analysis as novel biomarkers may appear in both sample types.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Kitzman, PhD, Principal Investigator — Baylor Scott & White Health and Wellness Center
Locations (1):
- Baylor Scott & White Health and Wellness Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Mendu ML, Erickson KF, Hostetter TH, Winkelmayer WC, Olan G, Meyer RN, Hakim R, Sedor JR. Federal Funding for Kidney Disease Research: A Missed Opportunity. Am J Public Health. 2016 Mar;106(3):406-7. doi: 10.2105/AJPH.2015.303009. No abstract available. PMID 26885959
- [Background] Saran R, Li Y, Robinson B, Abbott KC, Agodoa LY, Ayanian J, Bragg-Gresham J, Balkrishnan R, Chen JL, Cope E, Eggers PW, Gillen D, Gipson D, Hailpern SM, Hall YN, He K, Herman W, Heung M, Hirth RA, Hutton D, Jacobsen SJ, Kalantar-Zadeh K, Kovesdy CP, Lu Y, Molnar MZ, Morgenstern H, Nallamothu B, Nguyen DV, O'Hare AM, Plattner B, Pisoni R, Port FK, Rao P, Rhee CM, Sakhuja A, Schaubel DE, Selewski DT, Shahinian V, Sim JJ, Song P, Streja E, Kurella Tamura M, Tentori F, White S, Woodside K, Hirth RA. US Renal Data System 2015 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2016 Mar;67(3 Suppl 1):Svii, S1-305. doi: 10.1053/j.ajkd.2015.12.014. No abstract available. PMID 26925525
- [Background] Gargiulo R, Suhail F, Lerma EV. Cardiovascular disease and chronic kidney disease. Dis Mon. 2015 Sep;61(9):403-13. doi: 10.1016/j.disamonth.2015.07.005. Epub 2015 Aug 29. No abstract available. PMID 26328516
- [Background] Banks J, Marmot M, Oldfield Z, Smith JP. Disease and disadvantage in the United States and in England. JAMA. 2006 May 3;295(17):2037-45. doi: 10.1001/jama.295.17.2037. PMID 16670412
- [Background] So BH, Methven S, Hair MD, Jardine AG, MacGregor MS. Socio-economic status influences chronic kidney disease prevalence in primary care: a community-based cross-sectional analysis. Nephrol Dial Transplant. 2015 Jun;30(6):1010-7. doi: 10.1093/ndt/gfu408. Epub 2015 Jan 13. PMID 25586406
- [Background] Vart P, Gansevoort RT, Coresh J, Reijneveld SA, Bultmann U. Socioeconomic measures and CKD in the United States and The Netherlands. Clin J Am Soc Nephrol. 2013 Oct;8(10):1685-93. doi: 10.2215/CJN.12521212. Epub 2013 Jun 27. PMID 23813554
- [Background] Peralta CA, Vittinghoff E, Bansal N, Jacobs D Jr, Muntner P, Kestenbaum B, Lewis C, Siscovick D, Kramer H, Shlipak M, Bibbins-Domingo K. Trajectories of kidney function decline in young black and white adults with preserved GFR: results from the Coronary Artery Risk Development in Young Adults (CARDIA) study. Am J Kidney Dis. 2013 Aug;62(2):261-6. doi: 10.1053/j.ajkd.2013.01.012. Epub 2013 Mar 7. PMID 23473985
- [Background] Goraya N, Simoni J, Jo C, Wesson DE. Dietary acid reduction with fruits and vegetables or bicarbonate attenuates kidney injury in patients with a moderately reduced glomerular filtration rate due to hypertensive nephropathy. Kidney Int. 2012 Jan;81(1):86-93. doi: 10.1038/ki.2011.313. Epub 2011 Aug 31. PMID 21881553
- [Background] Goraya N, Simoni J, Jo CH, Wesson DE. A comparison of treating metabolic acidosis in CKD stage 4 hypertensive kidney disease with fruits and vegetables or sodium bicarbonate. Clin J Am Soc Nephrol. 2013 Mar;8(3):371-81. doi: 10.2215/CJN.02430312. Epub 2013 Feb 7. PMID 23393104
- [Background] Goraya N, Simoni J, Jo CH, Wesson DE. Treatment of metabolic acidosis in patients with stage 3 chronic kidney disease with fruits and vegetables or oral bicarbonate reduces urine angiotensinogen and preserves glomerular filtration rate. Kidney Int. 2014 Nov;86(5):1031-8. doi: 10.1038/ki.2014.83. Epub 2014 Apr 2. PMID 24694986
- [Background] Young BA, Katz R, Boulware LE, Kestenbaum B, de Boer IH, Wang W, Fulop T, Bansal N, Robinson-Cohen C, Griswold M, Powe NR, Himmelfarb J, Correa A. Risk Factors for Rapid Kidney Function Decline Among African Americans: The Jackson Heart Study (JHS). Am J Kidney Dis. 2016 Aug;68(2):229-239. doi: 10.1053/j.ajkd.2016.02.046. Epub 2016 Apr 9. PMID 27066930
- [Background] Boeing H, Bechthold A, Bub A, Ellinger S, Haller D, Kroke A, Leschik-Bonnet E, Muller MJ, Oberritter H, Schulze M, Stehle P, Watzl B. Critical review: vegetables and fruit in the prevention of chronic diseases. Eur J Nutr. 2012 Sep;51(6):637-63. doi: 10.1007/s00394-012-0380-y. Epub 2012 Jun 9. PMID 22684631
- [Background] Rehm CD, Penalvo JL, Afshin A, Mozaffarian D. Dietary Intake Among US Adults, 1999-2012. JAMA. 2016 Jun 21;315(23):2542-53. doi: 10.1001/jama.2016.7491. PMID 27327801
- [Background] Newgard CB. Metabolomics and Metabolic Diseases: Where Do We Stand? Cell Metab. 2017 Jan 10;25(1):43-56. doi: 10.1016/j.cmet.2016.09.018. Epub 2016 Oct 27. PMID 28094011
- [Background] Ganna A, Salihovic S, Sundstrom J, Broeckling CD, Hedman AK, Magnusson PK, Pedersen NL, Larsson A, Siegbahn A, Zilmer M, Prenni J, Arnlov J, Lind L, Fall T, Ingelsson E. Large-scale metabolomic profiling identifies novel biomarkers for incident coronary heart disease. PLoS Genet. 2014 Dec 11;10(12):e1004801. doi: 10.1371/journal.pgen.1004801. eCollection 2014 Dec. PMID 25502724
- [Background] Leaf DE, Jacob KA, Srivastava A, Chen ME, Christov M, Juppner H, Sabbisetti VS, Martin A, Wolf M, Waikar SS. Fibroblast Growth Factor 23 Levels Associate with AKI and Death in Critical Illness. J Am Soc Nephrol. 2017 Jun;28(6):1877-1885. doi: 10.1681/ASN.2016080836. Epub 2016 Dec 27. PMID 28028134
- [Background] Xue C, Yang B, Zhou C, Dai B, Liu Y, Mao Z, Yu S, Mei C. Fibroblast Growth Factor 23 Predicts All-Cause Mortality in a Dose-Response Fashion in Pre-Dialysis Patients with Chronic Kidney Disease. Am J Nephrol. 2017;45(2):149-159. doi: 10.1159/000454959. Epub 2016 Dec 23. PMID 28006765
- [Background] Rescigno T, Micolucci L, Tecce MF, Capasso A. Bioactive Nutrients and Nutrigenomics in Age-Related Diseases. Molecules. 2017 Jan 8;22(1):105. doi: 10.3390/molecules22010105. PMID 28075340
- [Background] Wilson DK, Kitzman-Ulrich H, Resnicow K, Van Horn ML, St George SM, Siceloff ER, Alia KA, McDaniel T, Heatley V, Huffman L, Coulon S, Prinz R. An overview of the Families Improving Together (FIT) for weight loss randomized controlled trial in African American families. Contemp Clin Trials. 2015 May;42:145-57. doi: 10.1016/j.cct.2015.03.009. Epub 2015 Mar 30. PMID 25835731
- [Background] Wilson DK, Kitzman-Ulrich H, Williams JE, Saunders R, Griffin S, Pate R, Van Horn ML, Evans A, Hutto B, Addy CL, Mixon G, Sisson SB. An overview of "The Active by Choice Today" (ACT) trial for increasing physical activity. Contemp Clin Trials. 2008 Jan;29(1):21-31. doi: 10.1016/j.cct.2007.07.001. Epub 2007 Jul 17. PMID 17716952
- [Background] Wilson DK, Trumpeter NN, St George SM, Coulon SM, Griffin S, Lee Van Horn M, Lawman HG, Wandersman A, Egan B, Forthofer M, Goodlett BD, Kitzman-Ulrich H, Gadson B. An overview of the "Positive Action for Today's Health" (PATH) trial for increasing walking in low income, ethnic minority communities. Contemp Clin Trials. 2010 Nov;31(6):624-33. doi: 10.1016/j.cct.2010.08.009. Epub 2010 Aug 27. PMID 20801233
- [Background] Kitzman H, Dodgen L, Mamun A, Slater JL, King G, Slater D, King A, Mandapati S, DeHaven M. Community-based participatory research to design a faith-enhanced diabetes prevention program: The Better Me Within randomized trial. Contemp Clin Trials. 2017 Nov;62:77-90. doi: 10.1016/j.cct.2017.08.003. Epub 2017 Aug 12. PMID 28807739
- [Background] Armstrong C; Joint National Committee. JNC8 guidelines for the management of hypertension in adults. Am Fam Physician. 2014 Oct 1;90(7):503-4. No abstract available. PMID 25369633
- [Background] Scialla JJ, Parekh RS, Eustace JA, Astor BC, Plantinga L, Jaar BG, Shafi T, Coresh J, Powe NR, Melamed ML. Race, Mineral Homeostasis and Mortality in Patients with End-Stage Renal Disease on Dialysis. Am J Nephrol. 2015;42(1):25-34. doi: 10.1159/000438999. Epub 2015 Aug 20. PMID 26287973
- [Background] Gutierrez OM, Rostand SG. Chronic kidney disease in African Americans: past, present, and future: introduction. Semin Nephrol. 2013 Sep;33(5):407-8. doi: 10.1016/j.semnephrol.2013.07.001. No abstract available. PMID 24119845
- [Background] Gutierrez OM, Parsa A, Isakova T, Scialla JJ, Chen J, Flack JM, Nessel LC, Gupta J, Bellovich KA, Steigerwalt S, Sondheimer JH, Wright JT Jr, Feldman HI, Kusek JW, Lash JP, Wolf M. Genetic African Ancestry and Markers of Mineral Metabolism in CKD. Clin J Am Soc Nephrol. 2016 Apr 7;11(4):653-62. doi: 10.2215/CJN.08020715. Epub 2016 Feb 8. PMID 26912553
- [Background] Gutierrez OM, Judd SE, Irvin MR, Zhi D, Limdi N, Palmer ND, Rich SS, Sale MM, Freedman BI. APOL1 nephropathy risk variants are associated with altered high-density lipoprotein profiles in African Americans. Nephrol Dial Transplant. 2016 Apr;31(4):602-8. doi: 10.1093/ndt/gfv229. Epub 2015 Jul 6. PMID 26152403
- [Background] Saneei P, Salehi-Abargouei A, Esmaillzadeh A, Azadbakht L. Influence of Dietary Approaches to Stop Hypertension (DASH) diet on blood pressure: a systematic review and meta-analysis on randomized controlled trials. Nutr Metab Cardiovasc Dis. 2014 Dec;24(12):1253-61. doi: 10.1016/j.numecd.2014.06.008. Epub 2014 Jun 27. PMID 25149893
- [Background] Breier M, Wahl S, Prehn C, Fugmann M, Ferrari U, Weise M, Banning F, Seissler J, Grallert H, Adamski J, Lechner A. Targeted metabolomics identifies reliable and stable metabolites in human serum and plasma samples. PLoS One. 2014 Feb 24;9(2):e89728. doi: 10.1371/journal.pone.0089728. eCollection 2014. PMID 24586991
- [Background] Carayol M, Licaj I, Achaintre D, Sacerdote C, Vineis P, Key TJ, Onland Moret NC, Scalbert A, Rinaldi S, Ferrari P. Reliability of Serum Metabolites over a Two-Year Period: A Targeted Metabolomic Approach in Fasting and Non-Fasting Samples from EPIC. PLoS One. 2015 Aug 14;10(8):e0135437. doi: 10.1371/journal.pone.0135437. eCollection 2015. PMID 26274920
- [Background] Nkuipou-Kenfack E, Duranton F, Gayrard N, Argiles A, Lundin U, Weinberger KM, Dakna M, Delles C, Mullen W, Husi H, Klein J, Koeck T, Zurbig P, Mischak H. Assessment of metabolomic and proteomic biomarkers in detection and prognosis of progression of renal function in chronic kidney disease. PLoS One. 2014 May 9;9(5):e96955. doi: 10.1371/journal.pone.0096955. eCollection 2014. PMID 24817014
- [Background] Dallmann G, Klavins K, Koal T. Targeted Quantitative Metabolomics Using Dried Plasma Spot Cards. https:novilytic.com/wp-content/uploads/2015/01/Metabolomics-with-Noviplex-Cards.pdf
- [Background] Hong DS, Oh IH, Park JS, Lee CH, Kang CM, Kim GH. Evaluation of Urinary Indices for Albuminuria and Proteinuria in Patients with Chronic Kidney Disease. Kidney Blood Press Res. 2016;41(3):258-66. doi: 10.1159/000443429. Epub 2016 Apr 29. PMID 27160690
- [Background] Thompson FE, Dixit-Joshi S, Potischman N, Dodd KW, Kirkpatrick SI, Kushi LH, Alexander GL, Coleman LA, Zimmerman TP, Sundaram ME, Clancy HA, Groesbeck M, Douglass D, George SM, Schap TE, Subar AF. Comparison of Interviewer-Administered and Automated Self-Administered 24-Hour Dietary Recalls in 3 Diverse Integrated Health Systems. Am J Epidemiol. 2015 Jun 15;181(12):970-8. doi: 10.1093/aje/kwu467. Epub 2015 May 10. PMID 25964261
- [Background] Institute Nc. ASA24 Automated Self-Administered 24-Hour Dietary Assessment Tool. http://epi.grants.cancer.gov/asa24/
- [Background] Glick HA, Doshi JA, Sonnad SS, Polsky D. Economic Evaluation in Clinical Trials. Oxford: Oxford University Press; 2007.
- [Background] Russell LB, Gold MR, Siegel JE, Daniels N, Weinstein MC. The role of cost-effectiveness analysis in health and medicine. Panel on Cost-Effectiveness in Health and Medicine. JAMA. 1996 Oct 9;276(14):1172-7. PMID 8827972